CLINICAL TRIAL: NCT07321912
Title: A Phase II Open Label Basket Trial Study Using Eflornithine (DFMO) for Ewing Sarcoma and Osteosarcoma
Brief Title: Eflornithine (DFMO) for Ewing Sarcoma and Osteosarcoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: USWM, LLC (dba US WorldMeds) (Industry)
Responsible Party: Principal Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCC023
Record Dates: First submitted 2026-01-05; First posted 2026-01-07 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Osteosarcoma; Ewing Sarcoma; Ewing Sarcoma Metastatic
MeSH Terms: conditions — Osteosarcoma; Sarcoma, Ewing | interventions — Eflornithine; Topotecan; Cyclophosphamide; Vincristine; Doxorubicin; Ifosfamide; Etoposide; Cisplatin; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Relapsed or Refractory Ewing Sarcoma Eligible to Receive Local Control (Experimental): DFMO will be administered as concurrent therapy during treatment of Ewing sarcoma. Participants completing treatment without experiencing an analytic event will continue to receive DFMO monotherapy as a maintenance treatment for an additional 24 months.
  Interventions: Drug: Eflornithine; Drug: Topotecan; Drug: Cyclophosphamide
- Cohort 2: Ewing Sarcoma Patients who are Metastatic at Diagnosis (Experimental): DFMO will be administered as concurrent therapy during consolidation treatment of metastatic Ewing sarcoma. Participants completing consolidation treatment without experiencing an analytic event will continue to receive DFMO monotherapy as a post consolidation maintenance treatment for an additional 24 months.
  Interventions: Drug: Eflornithine; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Doxorubicin; Drug: Ifosfamide; Drug: Etoposide
- Cohort 3: Osteosarcoma with relapse in the lung after resection of lung metastases (Experimental): DFMO will be dosed twice daily for 730 days.
  Interventions: Drug: Eflornithine
- Cohort 4A: Osteosarcoma with Poor Response to Induction Therapy at Completion of Local Control (Experimental): DFMO will be administered as concurrent therapy during Cycles 4-6 of post-surgery consolidation. Participants completing MAP without experiencing an analytic event will continue to receive DFMO monotherapy as a post consolidation maintenance treatment for an additional 24 months.
  Interventions: Drug: Eflornithine; Drug: Doxorubicin; Drug: Cisplatin; Drug: Methotrexate
- Cohort 4B: Osteosarcoma with Metastatic Disease at Diagnosis at Completion of Local Control (Experimental): DFMO will be administered as concurrent therapy during Cycles 4-6 of post-surgery consolidation. Participants completing MAP without experiencing an analytic event will continue to receive DFMO monotherapy as a post consolidation maintenance treatment for an additional 24 months.
  Interventions: Drug: Eflornithine; Drug: Doxorubicin; Drug: Cisplatin; Drug: Methotrexate

INTERVENTIONS:
Drug: Eflornithine — Oral twice daily
  Other Names: DFMO
Drug: Topotecan — IV
  Arms: Cohort 1: Relapsed or Refractory Ewing Sarcoma Eligible to Receive Local Control
Drug: Cyclophosphamide — IV
  Arms: Cohort 1: Relapsed or Refractory Ewing Sarcoma Eligible to Receive Local Control; Cohort 2: Ewing Sarcoma Patients who are Metastatic at Diagnosis
Drug: Vincristine — IV
  Arms: Cohort 2: Ewing Sarcoma Patients who are Metastatic at Diagnosis
Drug: Doxorubicin — IV
  Arms: Cohort 2: Ewing Sarcoma Patients who are Metastatic at Diagnosis; Cohort 4A: Osteosarcoma with Poor Response to Induction Therapy at Completion of Local Control; Cohort 4B: Osteosarcoma with Metastatic Disease at Diagnosis at Completion of Local Control
Drug: Ifosfamide — IV
  Arms: Cohort 2: Ewing Sarcoma Patients who are Metastatic at Diagnosis
Drug: Etoposide — IV
  Arms: Cohort 2: Ewing Sarcoma Patients who are Metastatic at Diagnosis
Drug: Cisplatin — IV
  Arms: Cohort 4A: Osteosarcoma with Poor Response to Induction Therapy at Completion of Local Control; Cohort 4B: Osteosarcoma with Metastatic Disease at Diagnosis at Completion of Local Control
Drug: Methotrexate — IV
  Arms: Cohort 4A: Osteosarcoma with Poor Response to Induction Therapy at Completion of Local Control; Cohort 4B: Osteosarcoma with Metastatic Disease at Diagnosis at Completion of Local Control

SUMMARY:
Ewing sarcoma (EWS) and osteosarcoma primarily affect adolescents and young adults. Common treatments include chemotherapy, surgery and radiation, however, there have been few recent advancements in the standard of care. By incorporating eflornithine (DFMO) as an additional therapy and/or maintenance therapy we hope to safely observe improved event-free survival and overall survival. There are 5 cohorts covered under this master protocol.

ELIGIBILITY:
Cohort 1:

Inclusion Criteria:

1. Participants must be ≤50 years of age at enrollment.
2. Histologically confirmed Ewing sarcoma that is refractory or in first or subsequent relapse. Histological confirmation either at initial diagnosis or disease progression.

   * Relapsed: Participants that have achieved CR at any point and then relapsed following/during standard of care therapy.
   * Refractory: Participants that failed to achieve CR after standard of care therapy or having progressed during standard of care therapy.
   * Note: Standard of care therapy for Ewing sarcoma includes multi-agent chemotherapy with local control consisting of either surgery and/or radiation therapy.
3. Extent of disease is judged by treating team to be amenable to the delivery of definitive local control (either definitive radiation, surgery, or a combination of these) at the time of study enrollment (to be completed after protocol defined Cycle 2).
4. Participants may enroll anytime during Cycle 1 or 2, prior to local control, as long as they received the same treatment during Cycle 1 and 2 as prescribed in this protocol.
5. Relapsed or refractory disease, including at least one of the following:

   * Tumor by CT or MRI
   * FDG-PET that is positive for disease
   * Bone Marrow biopsy/aspirate that is positive for disease

   Organ Function Requirements:
6. Participants must have adequate renal function as defined as:

   * For participants < 17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
   * For participants ≥17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Cockcroft and Gault formula (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Cockcroft and Gault formula is: [(140-age) x (Wt in kg) x (0.85 if female)] / (72 x SCr)
   * OR a 24 hour urine Creatinine clearance ≥ 70 mL/min/1.73 m2
7. Adequate liver function defined as:

   1. Total bilirubin ≤1.5 x upper limit of normal (ULN) for age, and
   2. SGPT (ALT <3 x upper limit of normal (ULN) for age (except for participants with liver metastasis who may enroll if ALT < 5 times ULN for age).
8. Adequate cardiac function defined as:

   1. Shortening fraction of ≥27% or
   2. Ejection fraction of ≥50%
9. Participants must have fully recovered from the hematological and bone marrow suppression effects of prior chemotherapy.
10. Participants must have a Lansky Play Scale or Karnofsky Performance Scale score of ≥ 60.
11. Participants of childbearing potential must have a negative pregnancy test and agree to use an effective birth control method. Participants who are lactating must agree to stop breast-feeding.
12. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all participants (or participants' legal representative).

Exclusion Criteria:

1. BSA of <0.25 m2
2. Participants with current CNS disease.
3. Investigational Drugs: Participants who are currently receiving another investigational drug are excluded from participation.
4. Anti-cancer Agents: Participants who are currently receiving other anticancer agents are not eligible.
5. Infection: Participants who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
6. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Cohort 2:

Inclusion Criteria:

* Age

  1. Participants must be ≤50 years of age at enrollment.

     Note:

     • Infants and small children are eligible for this study, however, the treating physicians and family must be prepared to deliver adequate local control as required in this study (see BCC Surgical and Imaging Guidelines).

     Diagnosis
  2. Participants with histologic diagnosis (by institutional pathologist) of newly diagnosed Ewing sarcoma or peripheral primitive neuroectodermal tumor (PNET) arising from bone or soft tissue and with metastatic disease involving lung, bone, bone marrow, or other metastatic site.

     For the purpose of this study, metastatic disease is defined as one or more of the following:
     * Lesions which are discontinuous from the primary tumor, are not regional lymph nodes, and do not share a bone or body cavity with the primary tumor. Skip lesions in the same bone as the primary tumor do not constitute metastatic disease. Skip lesions in an adjacent bone are considered bone metastases. If there is any doubt whether lesions are metastatic, a biopsy of those lesions should be performed.
     * Contralateral pleural effusion and/or contralateral pleural nodules.
     * Distant lymph node involvement.
     * Participants with pulmonary nodules are considered to have metastatic disease if the participant has:

       * Solitary nodule ≥0.5 cm or multiple nodules of ≥0.3 cm unless lesion is biopsied and negative for tumor;
       * Participants with solitary nodule <0.5 cm or multiple nodules <0.3 cm are not considered to have lung metastasis unless biopsy documents tumor.
     * Bone marrow metastatic disease is based on morphologic evidence of Ewing sarcoma based on H&E stains. In the absence of morphologic evidence of marrow involvement on H&E, participants with bone marrow involvement detected ONLY by flow cytometry, RT PCR, FISH, or immunohistochemistry will NOT be considered to have clinical bone marrow involvement for the purposes of this study.

     For participants that have a positive FDG-PET scan at study enrollment, a bilateral bone marrow biopsy will be required at study entry. If a bone marrow is required, the suggested approach for participants with large pelvic tumors in which a posterior iliac crest bone marrow biopsy would track through the tumor is to instead undergo 2 marrow biopsies on the contralateral side (either 2 posterior biopsies or one posterior and one anterior biopsy).

     • Bone metastasis: This study utilizes whole body FDG-PET scans to screen participants for bone metastases. Areas suspicious for bone metastasis based on FDG-PET scans require confirmatory anatomic imaging with either MRI or CT (whole body FDG-PET/CT or FDG-PET/MR scan acceptable). Whole body technetium bone scans may be performed at the discretion of the investigator and are not required. For participants without other sites of metastatic disease whose sole metastatic site to qualify for study entry is a single area suspicious for bone metastasis identified by FDG-PET, confirmatory biopsy or anatomic imaging evidence of an associated soft tissue mass at that site is required for study entry.

     Prior Therapy
  3. Participants must have completed 6 cycles of Induction therapy with VDC/IE per US standard of care (including standard modifications). Participants will enroll after the 6th cycle prior to local control.

     Organ Function Requirements
  4. Adequate renal function defined as:

     * For participants < 17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
     * For participants ≥17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Cockcroft and Gault formula (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Cockcroft and Gault formula is: [(140-age) x (Wt in kg) x (0.85 if female)] / (72 x SCr)
     * OR a 24 hour urine Creatinine clearance ≥ 70 mL/min/1.73 m2
  5. Adequate liver function defined as:

     * Total bilirubin ≤1.5 x upper limit of normal (ULN) for age, and
     * SGPT (ALT <3 x upper limit of normal (ULN) for age (except for participants with liver metastasis who may enroll if ALT < 5 times ULN for age).
  6. Adequate cardiac function defined as:

     * Shortening fraction of ≥27% or
     * Ejection fraction of ≥50%
  7. Participants must have fully recovered from the hematological and bone marrow suppression effects of prior chemotherapy.
  8. Participants must have a Lansky Play Scale or Karnofsky Performance Scale score of ≥ 60.
  9. Participants of childbearing potential must have a negative pregnancy test and agree to use an effective birth control method. Participants who are lactating must agree to stop breast-feeding.
  10. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all participants (or participants' legal representative).

Exclusion Criteria:

1. BSA of <0.25 m2
2. Investigational Drugs: Participants who are currently receiving another investigational drug are excluded from participation.
3. Anti-cancer Agents: Participants who are currently receiving other anticancer agents are not eligible.
4. Participants with regional node involvement as their only site of disease beyond the primary tumor.
5. Participants whose primary tumors arise in the intra-dural soft tissue (e.g. brain and spinal cord).
6. Participants with current CNS disease
7. Infection: Participants who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
8. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Cohort 3:

Inclusion Criteria:

* Age

  1. Participants must be less than 30 years of age at enrollment.

     Diagnosis
  2. Participants must have histologic diagnosis of osteosarcoma at original diagnosis.
  3. Participants must have had at least one episode of disease recurrence in the lungs without limitation on number of episodes of recurrence as long as they meet the following criteria:

     * Surgical resection of all possible sites of suspected pulmonary metastases in order to achieve a complete remission within 4 weeks prior to study enrollment*
     * Pathologic confirmation of metastases from at least one of the resected sites.
     * No local recurrence or metastatic disease elsewhere. *For participants with bilateral pulmonary metastases, resection must be performed from both lungs and the study enrollment must be within 4 weeks from date of the last lung surgery. No evidence of pulmonary metastatic disease; participants may have no visible lung nodules greater than 3 mm, and not considered to be disease.

     Note: If surgery related changes such as atelectasis are seen on the post-operative CT scan, participants will remain eligible to enroll as long as the operating surgeon believes that all sites of metastases were resected. Participants with positive microscopic margins will be eligible to enroll.

     Performance Level
  4. Participants must have a Lansky Play Scale or Karnofsky Performance Scale score of ≥ 60.

     Timing from Prior Therapy
  5. Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

     * Myelosuppressive anti-cancer therapy: Must not have been received within 2 weeks of study entry (4 weeks if prior nitrosourea).
     * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent.
     * Radiation therapy (RT): ≥2 weeks for local palliative RT (small port); ≥6 weeks must have elapsed if prior craniospinal RT or if ≥50% radiation of pelvis; ≥6 weeks must have elapsed if other substantial BM radiation.
     * Surgery: ≥2 weeks from last major surgery, including pulmonary metastasectomy, with the exclusion of a central line placement and core needle or small open biopsies.

     Organ Function Requirements
  6. Hematological:

     * Platelet count ≥50,000/μL without transfusion in last 7 days
     * Hgb ≥8.5 without transfusion in last 7 days
  7. Adequate renal function defined as:

     * For participants < 17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
     * For participants ≥17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Cockcroft and Gault formula (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Cockcroft and Gault formula is: [(140-age) x (Wt in kg) x (0.85 if female)] / (72 x SCr)
     * OR a 24 hour urine Creatinine clearance ≥ 70 mL/min/1.73 m2
  8. Adequate liver function defined as:

     * Total bilirubin ≤1.5 x upper limit of normal (ULN) for age.
     * SGPT (ALT <3 x upper limit of normal (ULN) for age.
  9. Adequate cardiac function defined as:

     * Shortening fraction of ≥27%, or
     * Ejection fraction of ≥50%.
  10. Adequate pulmonary function defined as:

      o No evidence of dyspnea at rest, no history of exercise intolerance, and a pulse oximetry >94%.
  11. Participants of childbearing potential must have a negative pregnancy test and agree to use an effective birth control method. Participants who are lactating must agree to stop breast-feeding.
  12. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all participants (or participants' legal representative).

Exclusion Criteria:

1. BSA of <0.25 m2
2. Investigational Drugs: Participants who are currently receiving another investigational drug are excluded from participation.
3. Anti-cancer Agents: Participants who are currently receiving other anticancer agents are not eligible.
4. Participants with distant bone metastases at original diagnosis or any subsequent relapse (participants with only skip lesions will be eligible).
5. Participants with concurrent local and pulmonary recurrence at the time of most recent episode of disease recurrence preceding enrollment.

   Note: participants who had local recurrence previously that has been treated and then presented with an isolated pulmonary recurrence and met the surgical resection criteria stated above will be eligible (see IC #3 above).
6. Participants with primary refractory disease with progression of the primary tumor on initial therapy.
7. Participants with other sites of extra-pulmonary metastases at the time of any episode of disease recurrence preceding enrollment.
8. Infection: Participants who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
9. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in who compliance is likely to be suboptimal.

Cohort 4A/B:

Inclusion Criteria:

Diagnosis Both Cohorts

1. Participants must have high grade osteosarcoma and received gross total resection prior to start of Cycle 3 MAP therapy. Participants with positive margins are eligible and may receive radiation therapy. This includes secondary malignancies.

   o Note: craniofacial osteosarcoma is NOT permitted.
2. The primary tumor was resectable after the initial 2 cycles of MAP chemotherapy.
3. Participants must have had a non-contrast chest CT and primary tumor site imaging consisting of an MRI or CT for optimal visualization of primary tumor site prior to local control. Physical scans and scan reports must be available to submit to BCC.

   Note: Two-view plain radiographs of the primary tumor site can be performed for participants who have a metallic prosthetic implant instead of CT or MRI if a significant metal artifact would occur by those imaging modalities;

   Cohort A only
4. Participant must have poor response to induction chemotherapy (those with 10% or more viable tumor remaining after surgery) and localized tumor.

   Cohort B only
5. Have an initial diagnosis of high-grade metastatic extremity or axial osteosarcoma resectable by the treating team.

   o Note: Metastatic pulmonary disease is defined as 3 or more lesions >5 mm or 1 lesion >1 cm or biopsy proven pulmonary metastatic disease if not meeting these radiographic criteria;
6. No definite progression of metastatic disease and no evidence of new metastatic disease.
7. Following definitive primary surgery, complete removal of all metastases or complete removal planned and deemed feasible.

   Non-Diagnostic Inclusion Criteria, Both Cohorts Age
8. Participants must be ≥5 years and ≤40 years on date of diagnostic biopsy. Performance Level
9. Participants must have a Lansky Play Scale or Karnofsky Performance Scale score of ≥ 60. Participants whose performance status is adversely affected by a pathologic fracture but who are able to undergo treatment are eligible.

   Prior Therapy
10. Participants must have completed standard induction therapy for initial diagnosis osteosarcoma (2 cycles [10weeks]) of MAP, Local control (surgery, assessment of histologic response), and a post-surgery 3rd cycle (5 weeks) of MAP. Participants will enroll after the 3rd cycle of MAP.

    Organ Function Requirements
11. Participants must have adequate renal function defined:

    * For participants < 17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Bedside Schwartz equation (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Bedside Schwartz equation is: [(0.413) X (Height in cm)] / SCr
    * For participants ≥17 years old: estimated Glomerular Filtration rate (eGFR) as calculated from the Cockcroft and Gault formula (in units of mL/min/1.73 m2) or via radioisotope GFR of ≥ 70 mL/min/1.73 m2. The Cockcroft and Gault formula is: [(140-age) x (Wt in kg) x (0.85 if female)] / (72 x SCr)
    * OR a 24 hour urine Creatinine clearance ≥ 70 mL/min/1.73 m2
12. Adequate cardiac function defined as:

    * Shortening fraction of ≥28%, or
    * Ejection fraction of ≥50%
13. Adequate liver function defined as:

    * Total bilirubin ≤1.5 x upper limit of normal (ULN) for age
    * SGPT (ALT <3 x upper limit of normal (ULN) for age.
14. Participants must have fully recovered from the hematological and bone marrow suppression effects of prior chemotherapy.
15. Participants of childbearing potential must have a negative pregnancy test and agree to use an effective birth control method. Participants who are lactating must agree to stop breast-feeding.
16. Written informed consent in accordance with institutional and FDA guidelines must be obtained from all participants (or participants' legal representative).

Exclusion Criteria:

1. BSA of <0.25 m2
2. Investigational Drugs: Participants who are currently receiving another investigational drug are excluded from participation.
3. Anti-cancer Agents: Participants who are currently receiving other anticancer agents are not eligible.
4. Infection: Participants who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
5. Participants who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in who compliance is likely to be suboptimal.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 406 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2031-04-01 (Estimated); Study Completion 2036-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Cohort 1 participants with relapse free survival (RFS) during study | 2 years plus 5 years follow up
  Cohort 1: To determine if relapse-free survival (RFS) in participants with relapsed or refractory Ewing sarcoma treated with multiagent chemotherapy is improved with the addition of DFMO as compared to historical outcomes of participants treated with the same multiagent chemotherapy without DFMO.
Number of Cohort 2 participants with event-free survival (EFS) during study | 2 years plus 5 years follow up
  Cohort 2: To determine if event-free survival (EFS) in participants with newly diagnosed metastatic Ewing sarcoma treated with multiagent chemotherapy is improved with the addition of DFMO as compared to historical outcomes of participants treated with the same multiagent chemotherapy without DFMO.
Cohort 3: Number of Cohort 3 participants at 12 months with disease control | 1 year plus 5 years follow up
  To determine the 12-month disease control rate (DCR) in participants with completely resected recurrent osteosarcoma treated with DFMO as compared to historical controls.
Cohort 4A: Number of Cohort 4A participants with event-free survival (EFS) during study | 2 years plus 5 years follow up
  Examine whether the addition of DFMO to post-operative chemotherapy with cisplatin, doxorubicin, and methotrexate (MAP) improves the event-free survival (EFS) for participants with osteosarcoma having localized disease with a poor histological response to 10 weeks of pre-operative chemotherapy.
Cohort 4B: Number of Cohort 4B participants with event-free survival (EFS) during study | 2 years plus 5 years follow up
  Examine whether the addition of DFMO to post-operative chemotherapy with cisplatin, doxorubicin, and methotrexate (MAP) improves the event-free survival (EFS) for participants with osteosarcoma with metastatic disease at diagnosis (Cohort 4B).

SECONDARY OUTCOMES:
Length of time that participants experience Overall Survival (OS) | 10 Years
  To compare overall survival in DFMO-treated participants versus historical controls.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 2 years
  To characterize safety and tolerability of DFMO plus multiagent chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle SaulnierSholler, MD, Study Chair — Penn State Health Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Beat Childhood Cancer Research Consortium website — http://research.beatcc.org/